CLINICAL TRIAL: NCT06947031
Title: Efficacy and Safety of the Minimed 780G® Advanced Hybrid Closed Loop System (AHCL) in Patients With Type 1 Diabetes Undergoing Surgery
Acronym: AHCL & surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Other Study IDs: FM-CIE-0085-25
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D); Surgery, Day
Keywords: Type 1 diabetes; Advanced Hybrid Closed Loop system; Time in range; surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- AHCL: AHCL users (Minimed 780G) undergoing elective and emergent surgical procedures during the study period.
  Interventions: Device: AHCL

INTERVENTIONS:
Device: AHCL — The downloaded data will be analyzed prior to the surgical procedure. In accordance with standard clinical practice, a TBR time-under-range % (<54 mg/dL) or TBR time-under-range % (<70 mg/dL) greater than 4% will be identified, and the target glucose will be increased by 10 mg/dL relative to the previously established value. This is intended to reduce the risk of perioperative hypoglycemia.

SUMMARY:
An analytical observational study based on a cohort of patients who received training at San Ignacio University Hospital. Glycemic control metrics were compared between the perioperative and postoperative periods and the preoperative period using a paired t test. Glycemic control metrics were compared between the preoperative, intraoperative, and postoperative periods using a paired t test. Finally, a subgroup analysis was performed based on the type of procedure, percentage of sensor use, and duration of diabetes.

DETAILED DESCRIPTION:
Patients using the Minimed 780G device who completed training and clinical follow-up in the Endocrinology Unit of San Ignacio University Hospital. Through the clinical follow-up established by the unit, patients must inform their physicians if they will be undergoing elective surgery or contact the medical team if they require emergency surgery during the recruitment period.

Data Collection Prior to the Surgical Procedure Once enrolled in the study, information about the surgical procedure will be collected, including the type of procedure and approximate duration. Patients will then be asked to upload their data for viewing on the Medtronic Carelink platform https://carelink.minimed.com/app/login. Glucose monitoring data from the 14 days prior to the surgical procedure will be downloaded from this platform for subsequent analysis.

Prior to the Surgical Procedure The downloaded data will be analyzed prior to the surgical procedure. According to standard clinical practice, a %TBR time under range (<54 mg/dL) or %TBR time under range (<70 mg/dL) greater than 4% will be identified, and the target glucose will be increased by 10 mg/dL relative to the previously established value. This is to reduce the risk of perioperative hypoglycemia.

Data Collection After the Surgical Procedure Once the surgical procedure is complete, data on glycemic control will be downloaded again during the surgical period and the following 14 days. The data will be analyzed according to the Consensus for CGM Metrics in Inpatient Clinical Trials published in 2023 in the Journal of Diabetes Science and Technology, presented later in the text. This consensus aims to identify the most important metrics to measure in CGM studies in patients in the hospital setting and recommend target values for these metrics (32).

Once the patient is discharged, they will be contacted to confirm information about the surgical procedure, such as type of anesthesia, duration of surgery, and postoperative complications, whether related to infectious processes or poor glycemic control.

Data Analysis

The specific metrics mentioned in the Consensus for Continuous Glucose Monitoring Metrics in Inpatient Clinical Trials (22) are described below:

ELIGIBILITY:
Inclusion Criteria:Patients older than 18 years AHCL (Minimed 780G) users undergoing elective and urgent surgery during the study period.

Exclusion Criteria:

Patients whose pump use was discontinued during the perioperative period. Pregnant patients. Patients without sensor data in the 2 weeks before and after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes users of AHCL undergoing elective and urgent surgery during the study period.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Time in range | Duration fo the surgery
  Time spent in the range of 100 - 180 mg/dl during the surgery

SECONDARY OUTCOMES:
Time below range | Duration fo the surgery
  To determine safety by the percentage of mean time below the 70 mg/dl range (TBR) in the perioperative period of surgical procedures.
THRH | Duration fo the surgery
  To investigate the association between 70-100mg/dl (time at high risk of hypoglycaemia, THRH) and TBR <54mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Gómez Medina, Endocrinologyst, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The availability of information is for academic purposes. It is at the discretion of the principal investigator.